CLINICAL TRIAL: NCT06845137
Title: Impact of Tactile-Kinesthetic Stimulation and Soft Tissue Manipulation on Blood Cortisol Levels in Preterm Neonates Admitted to Pediatric Care Settings: a Prospective Experimental Study
Brief Title: Impact of Tactile Kinesthetic Stimulation and Soft Tissue Manipulation on Cortisol in Preterm
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: faizan kashoo, PT (Other)
Collaborators: Galgotias University (Unknown)
Responsible Party: Sponsor-Investigator, faizan kashoo, PT, Lecturer, Majmaah University
Organization: Majmaah University (Other)
Allocation: Not Applicable | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SEC/SAHS/PHD/24/09
Record Dates: First submitted 2025-02-20; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Neonatal Disorder
Keywords: Neonates, Cortisol, Massage, Tactile Stimulation
MeSH Terms: conditions — Infant, Newborn, Diseases | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): In this study, preterm neonates in the experimental group received TKS and STM as part of their intervention. TKS involved the passive range of motion exercises for the neonates' joints, aiming to enhance mobility and stimulate neuromuscular responses. STM, on the other hand, incorporated various techniques such as gentle stroking, petrissage, and percussion, all of which were designed to improve circulation and facilitate pain management. Stroking techniques provided a soothing effect, while petrissage-through kneading and compression-helped in muscle relaxation and circulation enhancement. Percussion techniques further contributed to muscle stimulation and fluid movement, ultimately supporting physiological stability. These interventions promoted venous return to the heart, cleared lactic acid buildup, and facilitated increased oxygen delivery to tissues. The improved blood flow also triggered endorphin release, serving as a natural pain reliever, thereby reducing discomfort and enh
  Interventions: Other: Tactile-Kinesthetic Stimulation (TKS) and Soft Tissue Manipulation (STM)
- Standard Treatment (Active Comparator): The Neonate will receive all the nursing care plan as described in experimental except tactile and massage from the therapist.
  Interventions: Other: Standard Therapy

INTERVENTIONS:
Other: Tactile-Kinesthetic Stimulation (TKS) and Soft Tissue Manipulation (STM) — Tactile-Kinesthetic Stimulation (TKS): TKS involves the application of tactile (touch) and kinesthetic (movement) stimuli to various parts of the body. This technique aims to enhance sensory awareness and motor control. TKS can include gentle tapping, brushing, or vibration on the skin, joints, or muscles. The sensory input provided through TKS helps in proprioceptive feedback, which is essential for improving body awareness, coordination, and movement patterns. It is often used in neurological rehabilitation to facilitate neuromuscular re-education and in pediatric therapy to promote sensory integration.
  Soft Tissue Manipulation (STM): STM involves various manual techniques applied to the soft tissues of the body, including muscles, tendons, ligaments, and fascia. These techniques can range from gentle stretching and mobilization to deeper techniques such as myofascial release, trigger point therapy, and deep tissue massage. STM aims to alleviate muscle tension, improve flexibility,
  Arms: Experimental Group
Other: Standard Therapy — Nursing care for preterm neonates involves a higher level of monitoring and specialized support due to their underdeveloped physiological systems. Nurses focus on maintaining thermal regulation through incubators or radiant warmers to prevent hypothermia, as preterm infants are more vulnerable to temperature instability. Respiratory support is critical, often requiring continuous positive airway pressure (CPAP) or mechanical ventilation to assist with immature lungs. Nutritional support is provided through intravenous fluids or gavage feeding (tube feeding) if the infant is not yet able to breastfeed or bottle-feed. Nurses also monitor for complications such as hypoglycemia, infection, and jaundice and administer antibiotics, vitamin K, and eye prophylaxis as needed. Developmentally supportive care is emphasized, including minimizing sensory overload and encouraging kangaroo care (skin-to-skin contact) to support bonding, promote growth, and help regulate the neonate's heart rate, temp
  Arms: Standard Treatment

SUMMARY:
Effect of Soft tissue Therapy in managing Procedural Pain among neonates admitted to the neonatal intensive care unit. This study focuses on procedural pain management with the help of Soft tissue manipulation, which includes various techniques like stroking and petrissage manipulations.

DETAILED DESCRIPTION:
Preterm neonates are highly vulnerable to stress due to their immature physiological systems and exposure to intensive medical treatments. Elevated blood cortisol levels, a key indicator of stress, have been linked to negative neurodevelopmental and physiological outcomes. Tactile-Kinesthetic Stimulation (TKS) and Soft Tissue Manipulation (STM) are non-invasive therapeutic approaches that may help alleviate stress and support overall development in preterm infants. TKS and STM were chosen for their proven benefits in promoting neurodevelopment, stress reduction, and physiological stability in preterm neonates. Unlike pharmacological interventions, these non-invasive therapies enhance blood circulation, regulate cortisol levels, and improve autonomic function, fostering growth and early adaptation to extrauterine life without adverse effects. This prospective experimental study aims to assess the impact of TKS and STM on blood cortisol levels and pain in preterm neonates admitted to pediatric care units. The intervention group will receive TKS and STM. TKS includes passive range of motion for upper and lower limbs whereas STM includes effleurage/stroking, petrissage, frictional and percussive manipulations daily for 24 minutes over four consecutive days, while the control group will receive standard neonatal care without additional interventions. Blood samples for cortisol measurement will be collected on days 1 and 4. Secondary outcomes will include physiological parameters such as heart rate, oxygen saturation, and weight gain. Statistical analyses will compare baseline and post-intervention cortisol levels within and between groups. Trained staff nurse will measure blood cortisol using ELISA. Participants, statisticians, and outcome assessors remain blinded. ELISA ensures high reliability (intra-assay CV <10%) and validity (correlates strongly with gold-standard mass spectrometry). Blood cortisol levels in preterm neonates can be influenced by factors like gestational age, birth weight, medical interventions, pain, stress, feeding patterns, and NICU environment. To control variability, standardized stimulation protocols, consistent feeding schedules, minimal handling outside interventions and controlled ambient conditions (light, noise, temperature) were maintained, ensuring that observed cortisol changes were primarily due to the intervention We anticipate that preterm neonates receiving TKS and STM will exhibit a significant reduction in blood cortisol levels and pain compared to those in the control group, along with improvements in secondary outcomes. This study aims to generate evidence supporting the efficacy of TKS and STM in reducing stress biomarkers, ultimately promoting their integration into neonatal care protocols to enhance the developmental outcomes of preterm infants

ELIGIBILITY:
Inclusion Criteria:

1. Underwent medical procedures associated with procedural pain, such as venipuncture, heel pricks, or tracheal intubation.
2. Preterm neonates (28 to 36 weeks of gestation)
3. Stable Neonates

Exclusion Criteria:

1. Post-Surgical/operative cases
2. Infants with neurological conditions such as siezures etc.
3. Neonates/infants with congenital anomalies.
4. Neonates with extremely low birth weight

Ages: 0 Days to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-03-20 (Estimated); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in the cortisol level | 4 days after intervention
  In neonates, particularly preterm infants, blood cortisol levels are used to evaluate stress and adrenal function.
  High cortisol levels may indicate physiological stress, infection, or discomfort, whereas persistently low levels could suggest adrenal insufficiency or an immature stress response. [Time Frame: Baseline, 4 days after the intervention.
  Cortisol measurements were taken after four days to capture the cumulative physiological response to TKS and STM while minimizing acute fluctuations. Measuring after each session could reflect transient stress responses, whereas assessing only at the end might overlook early adaptive changes. This timing balances short-term hormonal variations with meaningful longitudinal effects on neonatal stress regulation

SECONDARY OUTCOMES:
Change in Neonatal Infant Pain Scale (NIPS) | 4 days after intervention
  The Neonatal Infant Pain Scale (NIPS) is a behavioral assessment tool applicable to both preterm and full-term infants. It has a total score of 7, categorized as follows: 0-2 signifies no pain, 3-4 indicates mild to moderate pain, and a score above 4 suggests severe pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital, Roorkee, Uttarakhand, India